CLINICAL TRIAL: NCT00713427
Title: A Multi-Center, Single Arm, Prospective Study of the WallFlex™ Biliary Partially-covered Stent for the Palliative Treatment of Malignant Bile Duct Obstruction
Brief Title: Study of the WallFlex™ Biliary Partially-covered Stent for the Palliative Treatment of Malignant Bile Duct Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-WALLFLEX-BIL-PALL-002; E7020
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2009-08

CONDITIONS: Biliary Strictures Caused by Malignant Neoplasms
Keywords: Biliary; Strictures; Malignant; Neoplasm; Palliation
MeSH Terms: conditions — Constriction, Pathologic; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WallFlex Stent (Other): All patients meeting eligibility criteria recieve the WallFlex™ Biliary Partially-Covered Stent, which has regulatory clearance in the areas in which the study is being conducted.
  Interventions: Device: WallFlex™ Biliary Partially-Covered Stent

INTERVENTIONS:
Device: WallFlex™ Biliary Partially-Covered Stent — Implantable metal biliary stent intended for use in the palliative treatment of biliary strictures produced by malignant neoplasms. The stent is partially covered with a polymer to reduce the potential for tumor ingrowth through the stent.

SUMMARY:
This is a a prospective study of the WallFlex™ Biliary Partially-covered Stent designed to collect data to support regulatory clearance by the FDA in the United States and to determine the functionality of the WallFlex™ Biliary Partially Covered Stent as a Palliative treatment for malignant bile duct obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Inoperable extrahepatic biliary obstruction by any malignant process
* Indicated for metal stent placement for palliative treatment of biliary stricture(s) produced by malignant neoplasms
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

* Participation in another invesitgational study within 90 days prior to date of patient consent.
* Strictures that cannot be dialated enough to pass the delivery system
* Perforation of any duct within the biliary tree
* Presence of any esophageal or duodenal stent
* Patients for whom endoscopic procedures are contraindicated
* Patients with known senesitivity to any components of the stent or delivery system
* Patients with active hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walsh, M.D., Study Director — Boston Scientific Corporation; Guido Costamagna, M.D., Principal Investigator — Università Cattolica del Sacro Cuore, Policlinico A. Gemelli
Locations (6):
- ULB Erasme Hospital, Brussels, Belgium
- Hopital Edouard Herriot, Lyon, Cedex 3, France
- EVK Krankenhaus der Universitat Dusseldorf, Düsseldorf, Germany
- Asian Institute of Gastroenterology, Hyderabaad, India
- Università Cattolica del Sacro Cuore, Rome, Italy
- Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam, AZ, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WallFlex Stent
Started | 70
Completed | 66
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: 70 patients were enrolled, of whom 69 received a stent and were evaluated for baseline characteristics.
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 69
Age, Continuous [Mean (Full Range); unit: years] | 68.6 [34 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Malignant cause of bile duct stricture [Count of Participants; unit: Participants]
  Pancreatic | 47
  Cholangiocarcinoma | 9
  Ampullary | 4
  Gallbladder | 3
  Metastases from colon | 2
  Primary liver cancer invading common bile duct | 1
  Metastases from esophageal | 1
  Metastases from lung | 1
  Metastases from breast | 1
Stricture location [Count of Participants; unit: Participants]
  Distal common bile duct | 46
  Mid common bile duct | 15
  Papilla | 6
  Proximal common bile duct | 2
Number of study stents placed [Number; unit: Stents] — A total of 71 stents were placed, as two of the study participants required two stents to be placed due to the length of their strictures.
  Stents
    number of 60mm x10mm stents placed | 54
    number of 40mm x 10mm stents placed | 13
    number of 80mm x10mm stents placed | 3
    number of 60mm x 8mm stents placed | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Recurrent Biliary Obstruction
Description: Defined as absence of recurrent biliary obstruction defined as absence of biliary symptoms. Biliary symptoms, included, but were not limited to jaundice, itching, right upper quadrant abdominal pain, nausea, vomiting, fever, and dark urine. Symptom assessment occurred during the Screening/Baseline period and at all follow-up time points.
Time Frame: Up to 6 months post treatment or prior to death, whichever came first
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 66
Participants | 62

2. Secondary Outcome: Number of Adverse Events Related to the Device and/or Procedure
Description: Number of adverse events (serious and non-serious) related to the device and/or procedure were collected following informed consent, treatment, and at all follow-up timepoints.
Time Frame: From time participant signs informed consent until time participant exits study (up to 6 months following stent placement)
Measure: Number; unit: related adverse events
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 69
related adverse events | 9

3. Secondary Outcome: Number of Participants With Technical Stent Placement Success
Description: Technical stent placement success defined as the ability to deploy the stent in satisfactory position across the stricture
Time Frame: Initial stent placement procedure
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 69
Participants | 68

4. Secondary Outcome: Number of Participants With Occurrence of Re-intervention
Description: A re-intervention is defined as any type of endoscopic, percutaneous, or surgical procedure to improve biliary drainage after insertion of the initial study stent. Re-intervention does not include a second WallFlex stent placement during the 7 days post initial placement as a second stent could have been placed due to misplacement or failure to cover the entire stricture.
Time Frame: Up to 6 months post-initial study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 66
Participants | 6

5. Secondary Outcome: Change in Biliary Obstruction Symptoms
Description: Incidence of symptoms of biliary obstruction
Time Frame: up to 6 months post-initial study treatment
Measure: Mean (Standard Deviation); unit: count of symptoms
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 29
count of symptoms | .62 (.98)

6. Secondary Outcome: Time to Recurrent Biliary Obstruction
Description: Biliary obstruction symptoms were collected at all follow-up visits post treatment and included but not limited to jaundice, itching, right upper quadrant abdominal pain, nausea, vomiting, fever, and dark urine. The time to recurrent biliary obstruction was recorded.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 66
days | 110 (63)

7. Secondary Outcome: Change in Bilirubin
Description: Bilirubin change at 1 month following stent placement as assessed against bilirubin at baseline.
Time Frame: 1 month following stent placement
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | WallFlex Stent
Number analyzed (Participants) | 66
mg/dL | -1.9 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse event data collected from the time the participant signed the informed consent until completion of the 6 month follow-up visit (occurring 6 months post-initial study treatment)
Description: Reported on Adverse Events (Serious and Non-serious) related to the device and/or procedure.
Arm/Group | WallFlex Stent
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 9/69
Other Adverse Events (participants affected / at risk) | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex Stent (N=69)
Recurrent Biliary Obstruction (Gastrointestinal disorders) | 4 (4)
Cholecystitis (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Right Upper Quadrant Pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days